CLINICAL TRIAL: NCT04821310
Title: AN EXPLORATORY, MULTICENTER, RANDOMIZED, DOUBLE BLIND STUDY OF CLINICAL OUTCOMES, TOLERABILITY, AND SAFETY OF 2 DOSES OF ORAL PANTOPRAZOLE IN PEDIATRIC PARTICIPANTS AGED 1 TO 11 YEARS AND 12 TO 17 YEARS WHO REQUIRE MAINTENANCE THERAPY FOR HEALED EROSIVE ESOPHAGITIS
Brief Title: Protonix Treatment of Maintenance of Healing in Pediatric Participants Aged 1-11 Years and 12-17 Years
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: B1791094; 2023-508770-28-00 (Registry Identifier: CTIS (EU))
Record Dates: First submitted 2021-03-26; First posted 2021-03-29 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Esophagitis
Keywords: Erosive; esophagitis
MeSH Terms: conditions — Esophagitis

STUDY DESIGN:
Intervention Model Description: randomized, double-blind
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm 1 Full Dose Pantoprazole and matching placebo (Active Comparator): Full Healing Dose of pantoprazole
  Interventions: Drug: Full dose Pantoprazole plus matching placebo
- Arm 2 Half Dose Pantoprazole and matching placebo (Active Comparator): Half Healing Dose of pantoprazole
  Interventions: Drug: Half Dose Pantoprazole plus matching placebo

INTERVENTIONS:
Drug: Full dose Pantoprazole plus matching placebo — Full healing dose of pantoprazole plus matching placebo
  Arms: Arm 1 Full Dose Pantoprazole and matching placebo
Drug: Half Dose Pantoprazole plus matching placebo — Half healing dose of pantoprazole plus matching placebo
  Arms: Arm 2 Half Dose Pantoprazole and matching placebo

SUMMARY:
The purpose of this study is to explore the outcomes, tolerability and safety of 2 different doses of oral pantoprazole (full healing dose, half healing dose), assigned based upon weight, for the maintenance of healing of erosive esophagitis in pediatric participants aged 1 to 17 years with endoscopically-confirmed, healed erosive esophagitis.

DETAILED DESCRIPTION:
Explore the outcomes, tolerability and safety of 2 different doses of oral pantoprazole (full healing dose, half healing dose), assigned based upon weight, for the maintenance of healing of erosive esophagitis in pediatric participants aged 1 to 17 years with endoscopically-confirmed, healed erosive esophagitis.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have a documented erosive lesion with an Los Angeles (LA) Grade of A to D prior to starting Proton Pump Inhibitor treatment:
* Capable of giving signed informed consent/assent
* Willingness and ability of the participant or parent/legal guardian to complete the eDiary
* Willing and able to comply with all scheduled visits, treatment plan, laboratory tests, lifestyle considerations, and other study procedures, including the use of the eDiary.
* Male and female participants aged 1 to 17 years.
* Minimum body weight 7 kilogram and weight at least at the 5th percentile per the Center for Disease Control standard age and weight chart, for the participant's age.
* To be considered a female of non childbearing potential, the participant must meet at least 1 of the following criteria :
* Premenarchal: The investigator (or other appropriate staff) must discuss the participant's premenarchal status with the participant and parent/legal guardian at office visits and during telephone contacts, as participants who achieve menarche during the study would no longer be considered "female participants of non childbearing potential" and must comply with the protocol requirements applicable to women of childbearing potential.

Exclusion Criteria:

* Previous administration of an investigational drug or vaccine within 30 days (or as determined by the local requirement) or 5 half-lives preceding the first dose of study intervention used in this study (whichever is longer).
* Children that may be at high risk from procedural sedation should be carefully evaluated. Participants with a history of complications during prior procedural sedation
* History or presence of upper gastrointestinal anatomic or motor disorders
* Family history of malignant hyperthermia
* Known hypersensitivity to any Proton Pump Inhibitor, including pantoprazole or to any substituted benzimidazole or to any of the excipients.
* Any disorder requiring chronic (daily) use of warfarin, heparin, other anticoagulants, methotrexate, atazanavir or nelfinavir, clopidogrel, or potent inhibitors or inducers of CYP2C19 (eg, phenytoin, sulfamethoxazole, valproic acid, carbamazepine, and griseofulvin).
* Serum creatine kinase levels >3 x upper limit of normal.
* Known history of human immunodeficiency virus or clinical manifestations of acquired immune deficiency syndrome.
* Active malignancy of any type, or history of a malignancy. Participants with a history of malignancies that have been surgically removed or eradicated by irradiation or chemotherapy and who have no evidence of recurrence for at least 5 years before Screening are acceptable.
* Diagnosed as having or has received treatment for esophageal, gastric, pyloric channel, or duodenal ulceration within 30 days before the Screening visit.
* Alanine aminotransferase or blood urea nitrogen >2.0 upper limit of normal or estimated creatinine >1.5 X upper limit of normal for age or any other laboratory abnormality considered by the Investigator to be clinically significant within 14 days before the Baseline Visit (Day 1).
* Other acute or chronic medical or psychiatric condition including recent (within the past year) or active suicidal ideation or behavior or laboratory abnormality that may increase the risk associated with study participation or study intervention administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the participant inappropriate for entry into this study.
* Has, in the Investigator's opinion, a serious chronic condition (eg, diabetes, epilepsy), which is either not stable or not well controlled and may interfere with the conduct of the study.
* Has any condition possibly affecting drug absorption (eg, gastrectomy).

Prior or Concomitant Therapy:

* Frequent, repeated use of oral or parenteral glucocorticoids (eg, prednisone, prednisolone, dexamethasone). Steroid inhalers and topical steroids may be used.
* Pregnant female participants; breastfeeding female participants.
* Is unwilling or unable to comply with the Lifestyle Considerations section

Ages: 1 Year to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 43 (Actual)
Dates: Start 2022-01-13 (Actual); Primary Completion 2025-12-16 (Actual); Study Completion 2025-12-16 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with endoscopically confirmed maintenance of healing of erosive esophagitis at Week 24, considering patients with excessive use of rescue medication as treatment failures | Week 24
  Endoscopically confirmed maintenance of healing of erosive esophagitis at Week 24.

SECONDARY OUTCOMES:
Number of Participants With Change From Baseline in Physical Examinations and Vital Signs | Baseline up to 36 weeks
  Safety and tolerability will be assessed by physical examinations, blood pressure, and pulse rate.
Incidence of Adverse Events (AEs) | Baseline up to 36 weeks
Number of Participants With Change From Baseline in Laboratory Tests Results | Baseline up to 36 weeks
  Safety and tolerability will be assessed by clinical laboratory measurements

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (28):
- United States (8):
  - Baptist/Wolfson's Children's Hospital, Jacksonville, Florida
  - Nemours Children's Health, Jacksonville, Jacksonville, Florida
  - University of Rochester, Rochester, New York
  - University of Rochester Medical Center Clinical Research Center, Rochester, New York
  - Board of Regents of the University of Wisconsin System, Madison, Wisconsin
  - UW Health E Terrace Dr Medical Center, Madison, Wisconsin
  - University Hospital and UW Health Clinics, Madison, Wisconsin
  - UW Health 2275 Deming Way Clinic, Middleton, Wisconsin
- University clinical center of the Republic of Srpska, Banja Luka, Bosnia and Herzegovina
- Georgia (4):
  - JSC Georgian Clinics, Tbilisi
  - LTD Imedi Clinic, Tbilisi
  - Georgian-American Family Medicine Clinic, Tbilisi
  - Evex clinic after I. Tsitsishvili, Tbilisi
- India (2):
  - SR Kalla Memorial Gastro & General Hospital, Jaipur, Rajasthan
  - Medical college and Hospital, Kolkata, West Bengal
- Puerto Rico (2):
  - Hospital HIMA San Pablo Caguas, Caguas
  - Chiara Biaggi de Casenave, MD, Guaynabo
- Serbia (2):
  - University Children's Hospital, Belgrade
  - University Clinical Center of Kragujevac, Kragujevac
- Slovakia (2):
  - Univerzitna nemocnica Martin, Klinika deti a dorastu, Martin
  - KM Management, spol. s r.o.,, Nitra
- Turkey (Türkiye) (3):
  - MDX Klinik Arastirma Egitim ve Danismanlik Ltd, Istanbul
  - Izmir Saglik Bilimleri University Tepecik Training And Research Hospital, Izmir
  - T.C. Saglik Bakanligi - Izmir Sehir Hastanesi, Izmir
- United Kingdom (4):
  - Evelina London Children's Hospital, London
  - Guys & St Thomas Nhs Foundation, London
  - King's College Hospital NHS Foundation Trust, London
  - Great Ormond Street Hospital For Children NHS Foundation Trust, London

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=B1791094